CLINICAL TRIAL: NCT01911026
Title: The Impact of Nurse Education on the Quality of Inpatient Bowel Preparation for Colonoscopy; Randomized Single Blinded Study
Brief Title: The Impact of Nurse Education on the Quality of Inpatient Bowel Preparation for Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Kim Eun Soo, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-05-049-001
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Ottawa Scale <6
Keywords: Bowel preparation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Experimental): The investigational, or experimental arm, will receive standard written instructions on preparing for a colonoscopy plus interventional instructions from reinforcement educated nurse such as 'Reinforcement Nurse Education'
  Interventions: Other: Reinforcement Nurse Education
- Standard preparation instructions (No Intervention): The control arm will receive written instructions on preparing for a colonoscopy per standard of care at Keimyung University Dongsan Medical Center

INTERVENTIONS:
Other: Reinforcement Nurse Education — The investigational, or experimental arm, will receive standard written instructions on preparing for a colonoscopy plus instructions from reinforcement educated nurse
  Arms: Interventional

SUMMARY:
Effective bowel preparation is important for examination of the entire colon adequately and for identifying colonic lesions during colonoscopy. However, it is well known that bowel preparation of inpatients is much poorer than that of outpatients. Our goal is to improve bowel preparations with reinforcement of nurse education that explains the steps required for bowel preparation for inpatients undergoing colonoscopies. The education will focus on explaining the purpose of a screening colonoscopy, the rationale for bowel preparation, the pre-colonoscopy diet, and the instructions for completing the laxative. Patients in the control group will receive the standard written bowel preparation instructions, while patients in the intervention group will receive standard written instructions plus a explanation from reinforcement-educated nurse. The investigators hypothesize that patients received a explanation from reinforcement-educated nurses will lead to improved patient compliance and a better bowel preparation. In addition, the investigators hypothesize that a better quality bowel preparation will improve detection of colonic polyps and patients' satisfaction for colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* all inpatients
* age >18
* referred and scheduled for an elective screening colonoscopy

Exclusion Criteria:

* outpatients
* pregnancy
* breast feeding
* prior history of surgical large bowel resection
* patients allergic to PEG-ELS based laxatives

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | day 1
  The primary outcome will be the endoscopist's assessment of the quality of preparation using Boston and Ottawa bowel preparation scale

SECONDARY OUTCOMES:
Patient compliance | baseline
  Patient compliance with preparation instructions self-reported in a pre-procedure questionnaire
Colonoscope insertion and withdrawal times | day 1
  Time from insertion to cecum and time from cecum to anus
Patient's willingness to do bowel preparation next time | baseline
  Patient's willingness to do bowel preparation next time self-reported on a pre-procedure questionnaire
Preparation associated side effects | baseline
  Presence and severity of preparation associated side effects including: bloating, abdominal pain, and nausea/vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, Professor, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Eun Soo Kim, Daegu, South Korea